CLINICAL TRIAL: NCT04144218
Title: International Multicenter, Double-blind, Randomized, Placebo-controlled Evaluation of the Efficacy and Safety of Lacosamide in the Treatment of Pediatric Patients With Focal Refractory Epilepsy.
Brief Title: Evaluation of the Efficacy and Safety of Lacosamide in Pediatric Patients With Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Tongji Hospital (Other); Michigan State University (Other); Juntendo University (Other); Technical University of Munich (Other); RIKEN (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR20191016
Record Dates: First submitted 2019-10-17; First posted 2019-10-30 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet
- Experimental group (Experimental)
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — The experimental group will be given oral lacosamide supplementation on the basis of the original antiepileptic drugs.
  Arms: Experimental group
Drug: Placebo oral tablet — The control group will be given oral placebo supplementation on the basis of the original antiepileptic drugs.
  Arms: Control group

SUMMARY:
Children with focal refractory epilepsy will be routinely included in the collection of history, blood routine, biochemistry, EEG, MRI and 18F-FDG PET to determine the location of the epileptogenic focus and to assess the severity of the disease. This international multicenter clinical trial uses a double-blind, randomized, controlled study to evaluate the safety and efficacy of LCM in clinical applications in children with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of focal epilepsy with or without generalized seizures according to the 2017 International Association of Anti-Epilepsy (ILAE) classification criteria.
* Stable taking 1 or 2 other first-line anti-epileptic drugs for at least 10 weeks before screening visits.
* Seizure occurred during the 8-week retrospective baseline period with a complete medical record diary.

Exclusion Criteria:

* A history of status epilepticus within 3 months prior to screening visits.
* Poor adherence to previous treatment.
* Other serious organic diseases, mental illnesses and neurological diseases.
* Abnormal liver and kidney function and blood routine results.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-11-08 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of weekly seizures (times/week) | 16-week
  The reduction of absolute number of weekly seizures in the 16-week treatment period compared with the retrospective baseline period
Assessment of liver function by serum alanine aminotransferase (U/L) | One year
  The serum alanine aminotransferase (blood biochemistry) will be performed at baseline, at the 3rd and 6th visits to monitor the liver function of patients.
Assessment of renal function by serum creatinine (umol/L) | One year
  The serum creatinine (blood biochemistry) will be performed at baseline, at the 3rd and 6th visits to monitor the renal function of patients.
Assessment of white blood cell count ( /L) | One year
  The white blood cell count (blood routine) will be performed at baseline, at the 3rd and 6th visits to monitor the renal function of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine and PET/CT Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No